CLINICAL TRIAL: NCT02721810
Title: Engaging Surrogates and Physicians to Ensure Concordant Critical Care
Brief Title: Patient Engagement Initiative
Acronym: PEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00082272
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Prompts standard to rounds or electronic medical records.
- Prompting Intervention (Experimental): Prompting consideration of 3-month functional outcome.
  Interventions: Behavioral: Consideration of 3-month functional prognosis

INTERVENTIONS:
Behavioral: Consideration of 3-month functional prognosis
  Arms: Prompting Intervention

SUMMARY:
A no-cost intervention may improve adherence with a recommendation for higher-quality, lower-cost care for patients with critical illness endorsed by a collaborative of critical care societies. The investigators propose prompting consideration of functional outcomes. This trial will help establish the impact of the intervention on practice patterns including proxy engagement and elements of shared decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Licensed physicians
* At least 4 weeks of clinical work in an I.C.U. in the U.S.A. during the past 12 months

Exclusion Criteria:

* <25 years old
* Non-English speaking
* Primarily practicing medicine outside the U.S.A.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Presence of acceptable treatment option as assessed by a checklist completed by clinical colleges. | 0 to 5 minutes after prompting an intervention

SECONDARY OUTCOMES:
Level of conflict with proxy with a previously validated single question | 0 to 5 minutes after prompting an intervention
Level of shared decision-making measured using CollaboRATE scale | 0 to 5 minutes after prompting an intervention
Prevalence of communication skills for involving ICU proxies in treatment decisions assessed by a checklist completed by clinical colleges | 0 to 5 minutes after prompting an intervention
Medical interactions assessed using the Roter Interaction Analysis System (RIAS) | 0 to 5 minutes after prompting an intervention
Prevalence of the discussed option of stopping life support as assessed by blinded assessors | 0 to 5 minutes after prompting an intervention
Prevalence of conveying prognosis as assessed by blinded assessors | 0 to 5 minutes after prompting an intervention
Level of shared decision-making measured using CollaboRATE scale as assessed by blinded assessors | 0 to 5 minutes after prompting an intervention
The Observer OPTIONS5 measure completed by blinded assessors | 0 to 5 minutes after prompting an intervention
Consulting services requested by study participants | 0 to 5 minutes after prompting an intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Turnbull, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abshire MA, Li X, Basyal PS, Teply ML, Singh AL, Hayes MM, Turnbull AE. Actor feedback and rigorous monitoring: Essential quality assurance tools for testing behavioral interventions with simulation. PLoS One. 2020 May 29;15(5):e0233538. doi: 10.1371/journal.pone.0233538. eCollection 2020. PMID 32469920
- [Derived] Turnbull AE, Hayes MM, Brower RG, Colantuoni E, Basyal PS, White DB, Curtis JR, Needham DM. Effect of Documenting Prognosis on the Information Provided to ICU Proxies: A Randomized Trial. Crit Care Med. 2019 Jun;47(6):757-764. doi: 10.1097/CCM.0000000000003731. PMID 30882479